CLINICAL TRIAL: NCT06814678
Title: Effectiveness of Interactive Exergaming Combined With the Otago Exercise Program on Mobility in Older Individuals Living in Communities: A Cluster-Randomized Controlled Study
Brief Title: Interactive Exergaming With Otago Exercise Program on Mobility in Community-Dwelling Older Adults
Acronym: GAME-OEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, JIA-JING SUN, PhD Candidate, Registered Nurse, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202412HM008; Taiwan Nurses Association (Other Grant/Funding Number: TWNA-1141004)
Record Dates: First submitted 2025-01-24; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Physical Functional Performance; Psychological Health; Physical Fitness; Mobility Limitation; Aging
Keywords: Otago Exercise Program; Interactive exergaming; Mobility decline; Community-dwelling older adults; Physical performance; Intrinsic capacity; Psychological health; Muscle strength
MeSH Terms: conditions — Psychological Well-Being; Mobility Limitation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This cluster-randomized controlled trial uses parallel assignment where community centers are randomly allocated to either receive interactive exergaming combined with Otago Exercise Program intervention or usual care control group. All eligible participants within each cluster follow the same intervention protocol
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor who performs all measurements and evaluations will be blinded to group allocation throughout the study period. This assessor will not be involved in intervention delivery or have any contact with participants during exercise sessions to maintain masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group with Usual Care (Placebo Comparator): Participants in the control group will maintain their usual daily activities and routine care without any specific exercise intervention during the 12-week study period. They will receive standard health education materials and regular check-ups but no structured exercise program
  Interventions: Other: Control Group with Usual Care
- Interactive Exergaming with Otago Exercise Program (Experimental): A 12-week structured program consisting of 120 minutes per week divided into two 60-minute sessions. Each session combines Otago Exercise Program for strength and balance with interactive exergaming activities, conducted in community centers under certified instructor supervision with standardized equipment. Exercise intensity progresses according to individual performance.
  Interventions: Behavioral: Interactive Exergaming with Otago Exercise Program

INTERVENTIONS:
Behavioral: Interactive Exergaming with Otago Exercise Program — Participants will receive a 12-week structured program combining interactive exergaming and Otago Exercise Program. Sessions include balance training, strength exercises, and functional mobility activities delivered through interactive gaming platforms, supervised by trained instructors.
  Arms: Interactive Exergaming with Otago Exercise Program
Other: Control Group with Usual Care — Participants will maintain their regular activities at community centers or facilities, including cognitive therapy, oral exercises, and upper limb training programs, during the 12-week study period
  Arms: Control Group with Usual Care

SUMMARY:
This clinical trial aims to evaluate the effectiveness of interactive exergaming combined with Otago Exercise Program on mobility among community-dwelling older adults aged 65 and above. The main research questions are:

Does this combined exercise intervention improve elderly mobility? Does this program enhance muscle strength and psychological well-being?

Researchers will compare two groups: one group will do the combined exercise program for 12 weeks, while the other group will continue their usual activities.

Participants will:

* Have their health checked three times: at the start, after 12 weeks, and 3 months later
* If in the exercise group, attend exercise sessions twice a week for 12 weeks
* Complete tests about their physical abilities and how they feel emotionally

Who can take part:

* Adults age 65 or older
* People who need more than 12 seconds to stand up and sit down 5 times
* People who can stand for at least 30 seconds with support

People cannot take part if they have serious vision problems, recent leg injuries, major illnesses, significant memory problems, or mental health conditions.

DETAILED DESCRIPTION:
This cluster-randomized controlled trial investigates the integration of interactive exergaming with the evidence-based Otago Exercise Program (OEP) to enhance mobility among community-dwelling older adults. The study employs comprehensive methodology and rigorous assessment protocols to evaluate intervention effectiveness.

Methodology and Technical Implementation:

Assessment Tools and Measurements:

Primary Outcome Measures:

ICOPE (Integrated Care for Older People) screening tool evaluating six domains: cognition, mobility, nutrition, vision, hearing, and depression

Short Physical Performance Battery (SPPB, ICC=0.81-0.91) measuring:

Balance (side-by-side, semi-tandem, tandem stance) Gait speed (3-meter walk test) Lower extremity strength (5-time sit-to-stand)

Lower extremity muscle strength assessment using MicroFET2 digital dynamometer (accuracy ±1%):

Quadriceps strength Ankle dorsiflexion Hip abduction

Secondary Outcome Measures:

Three-Item Loneliness Scale (T-ILS, Cronbach's α=0.87) Geriatric Depression Scale-5 (GDS-5) Well-being Scale for Older Adults (9 items, Cronbach's α=0.91)

Intervention Protocol Design:

Exercise Program Structure:

12-week intervention period Two 60-minute sessions per week (120 minutes total) Group format (10-25 participants) Led by certified OEP trainers Integration of Nex Playground exergaming system

Session Components:

1. Warm-up (10 minutes):

   Head and neck rotations Back stretches Upper body rotation Lower limb stretches
2. Otago Exercise Program (30 minutes):

   Knee lifts Ankle movements Knee extensions Standing exercises with support Heel-toe exercises Sit-to-stand practice
3. Interactive Exergaming (20 minutes):

   Virtual soccer targeting lower limb strength Fruit Ninja for upper body engagement Alternating activities to prevent fatigue
4. Cool-down (10 minutes):

   Stretching exercises Relaxation techniques

   Technical Implementation:

   Equipment and Setting:

   Spacious, well-ventilated rooms Sturdy chairs with armrests Nex Playground gaming system Large display screen/projector Non-slip exercise mats Safety rails/supports

   Safety Protocols:

   Environmental risk assessment Fall prevention measures Emergency response procedures Continuous monitoring by trained staff Regular equipment maintenance

   Quality Control Measures:

   Standardization:

   Assessor training (ICC > 0.80 required) Intervention delivery protocols Documentation procedures Data collection methods

   Blinding:

   Outcome assessors blinded to group allocation Separate staff for intervention and assessment Data coding for anonymity

   Monitoring:

   Attendance tracking Adverse event documentation Intervention fidelity checks Regular team meetings

   Statistical Analysis Framework:

   Primary Analysis:

   Intention-to-treat principle Generalized Estimating Equations (GEE) Repeated measures analysis Cluster-level adjustments

   Data Management:

   Coded data entry Regular quality checks Missing data protocols Interim analyses

   Methodological Considerations:

   Cluster Randomization:

   Unit of randomization: community centers Stratification by center size Baseline characteristic balance Intraclass correlation adjustment

   Potential Challenges:

   Participant adherence Technology acceptance Health status changes Environmental factors Measurement biases

   Risk Mitigation:

   Regular communication Technical support Flexible scheduling Safety monitoring Modified exercises when needed

   Innovation and Scientific Contribution:

   This study offers several innovative aspects:

   Integration of traditional exercise with modern technology Comprehensive assessment of physical and psychological outcomes Rigorous methodology in community settings Focus on functional mobility and engagement Potential for scalability and sustainability

   The protocol addresses key challenges in elderly exercise programs by:

   Enhancing engagement through interactive technology Maintaining safety with structured progression Providing social interaction opportunities Enabling objective measurement of outcomes Supporting long-term adherence

   This research contributes to the field by:

   Evaluating a novel intervention approach Generating evidence for technology-enhanced exercise Addressing both physical and psychological outcomes Providing implementation guidance for community programs Supporting active aging initiatives

   The study's comprehensive approach and rigorous methodology aim to provide valuable evidence for improving mobility interventions in community-dwelling older adults, with potential implications for public health policy and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Abnormal mobility based on ICOPE screening (Five-time chair stand test > 12 seconds)
* Able to stand holding handrail for > 30 seconds

Exclusion Criteria:

* Severe visual impairment
* Lower limb fracture
* Acute serious illness
* Moderate to severe cognitive impairment (SPMSQ > 5 errors)
* Diagnosed psychiatric disorders

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-11 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mobility Performance | Baseline, 12 weeks, 3 months
  Measured by Short Physical Performance Battery (SPPB) Scale: 0-12 points, higher scores indicate better performance
Lower Extremity Strength | Baseline, 12 weeks, 3 months
  Measured by digital dynamometer Unit: Kilograms (kg)

SECONDARY OUTCOMES:
Intrinsic Capacity Score | baseline (T0), post 12-week intervention (T1), and 3-month follow-up (T2)
  omprehensive assessment of intrinsic capacity using Integrated Care for Older People (ICOPE) screening tool, measuring six domains:
  * Cognition (3 memory items and orientation questions)
  * Mobility (5-time sit-to-stand test)
  * Nutrition (weight loss and appetite assessment)
  * Vision (visual assessment)
  * Hearing (whisper test)
  * Depression (mood and interest assessment) For each domain, if any item within that domain is abnormal, the domain is scored as 0 (indicating risk of capacity decline); if all items are normal, the domain is scored as 1 (normal). Total score ranges from 0 (all domains at risk) to 6 (all domains normal), with higher scores indicating fewer domains at risk of capacity decline.
Loneliness Level | Measured at baseline (T0), post 12-week intervention (T1), and 3-month follow-up (T2)
  Three-Item Loneliness Scale (T-ILS) Assessment of loneliness using T-ILS. Scale: 3-9 points, lower scores indicate less loneliness
Depression Symptoms | Measured at baseline (T0), post 12-week intervention (T1), and 3-month follow-up (T2)
  Assessment of depression symptoms using Geriatric Depression Scale-5 (GDS-5). Scale: 0-5 points, lower scores indicate less depressive symptoms
Well-being Status | Measured at baseline (T0), post 12-week intervention (T1), and 3-month follow-up (T2)
  Assessment of well-being using 9-item Well-being Scale. Scale: 9-45 points, higher scores indicate better well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 105, Yusheng Street, Shilin District, Taipei City 111, Taiwan, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Protection of participant privacy and confidentiality. Institutional policies and ethical review board requirements.